CLINICAL TRIAL: NCT04244981
Title: Efficacy of Prothrombin Complex Concentrate Reducing Perioperative Blood Loss in Cardiac Surgery, Compared With Fresh Frozen Plasma: Study Protocol for a Non-inferiority, Randomized Controlled Trial
Brief Title: Efficacy of Prothrombin Complex Concentrate Reducing Perioperative Blood Loss in Cardiac Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: SHI Jia (Other)
Collaborators: Peking Union Medical College Hospital (Other); Beijing Anzhen Hospital (Other); Guizhou Provincial People's Hospital (Other); Zunyi Medical College (Other); First Affiliated Hospital of Harbin Medical University (Other); The First Affiliated Hospital of Air Force Medicial University (Other); The Affiliated Hospital Of Guizhou Medical University (Other)
Responsible Party: Sponsor-Investigator, SHI Jia, Vice Chair, the department of Anesthesiology, Chinese Academy of Medical Sciences, Fuwai Hospital
Organization: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PCC vs FFP Study
Record Dates: First submitted 2020-01-05; First posted 2020-01-28 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Cardiac Surgical Procedures
Keywords: prothrombin complex concentrate; fresh frozen plasma; perioperative blood loss; efficacy; cardiac surgery; cardiopulmonary bypass
MeSH Terms: conditions — Hemophilia B | interventions — Factor IX

STUDY DESIGN:
Intervention Model Description: 816 patients who meet the criteria will be randomly divided into 2 groups, named prothrombin complex concentrate group (group PCC) and fresh frozen plasma group (control group, group FFP), with 408 cases in each group. Preoperative management, anesthetic and surgical techniques will be standardized for all patients. Prolonged APTT (> 45 s) will be regarded as a trigger for administration of PCC or FFP, according to the randomized groups. In group PCC, patients will be given 8~15 IU/kg PCC. In group FFP, patients will be given 6~10 mL/kg FFP.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Allocation will be concealed using an interactive web response system, and nurse anaesthetists will prepare the corresponding products for each patient according to the group assignments in an anaesthesia preparation room. PCC or FFP will be pumped into 50 ml syringes firstly, covered with opaque paper to hide the contents. For group PCC, we first diluted PCC to 50ml with normal saline, and then supplemented subsequent volume using normal saline to make it equal to the corresponding required volume of FFP.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- PCC group (Experimental): When APTT is prolonged (> 45 s) measured 20 minutes after CPB or excessive bleeding observed, patients will be given 8～15 IU/kg PCC.
  Interventions: Drug: Prothrombin Complex Concentrate, Human
- FFP group (Active Comparator): When APTT is prolonged (> 45 s) measured 20 minutes after CPB or excessive bleeding observed, patients will be given 6～10 mL/kg FFP.
  Interventions: Drug: Fresh Frozen Plasma

INTERVENTIONS:
Drug: Prothrombin Complex Concentrate, Human — Four types of 4-factor prothrombin complex concentrate will be used.
  1. Human Prothrombin Complex (Rongsheng Pharmaceuticals Co., Ltd.), containing 300 IU factor IX, 300 IU factor II, 120 IU factor VII, and 300 IU factor X each bottle.
  2. Human Prothrombin Complex (China Resources Boya Biopharmaceutical Group Co., Ltd.), containing 400 IU factor IX, 400 IU factor II, 200 IU factor VII, and 400 IU factor X each bottle.
  3. Human Prothrombin Complex (Hualan Biological Engineering, INC.), containing 300 IU factor IX, 300 IU factor II, 75 IU factor VII, and 300 IU factor X each bottle.
  4. Human Prothrombin Complex (Shandong Taibang Biological Products Co., Ltd.), containing 300 IU factor IX, 300 IU factor II, 210 IU factor VII, and 300 IU factor X each bottle.
  When APTT is prolonged (> 45 s) measured 20 minutes after CPB or excessive bleeding observed, patients will be given 8～15 IU/kg PCC.
  Arms: PCC group
Drug: Fresh Frozen Plasma — When APTT is prolonged (> 45 s) measured 20 minutes after CPB or excessive bleeding observed, patients will be given 6～10 mL/kg FFP.
  Arms: FFP group

SUMMARY:
This study is a non-inferiority, randomized controlled trial, based on the hypothesis that 4-factor PCC is not inferior to FFP in reducing perioperative blood loss in patients undergoing cardiac surgery under cardiopulmonary bypass. 816 subjects will be randomly divided into 2 groups (group PCC and group FFP), with 408 cases in each group. Patients will be given 8~15 IU/kg 4-factor PCC in group PCC and 6~10 ml/kg FFP in group FFP. All the patients will be followed up respectively at 24 hours, 48 hours, 72 hours and 7 days after the surgery. The primary outcome is the volume of blood loss within 24 hours after surgery. The secondary outcomes include (1) the total units of allogeneic red blood cells (RBCs) transfused within 7 days after surgery and (2) hemostatic response (effective if no hemostatic interventions occurred from 60 minutes to 24 hours after treatment initiation). Adverse events and serious adverse events will be monitored as safety outcomes.

DETAILED DESCRIPTION:
Perioperative blood loss and allogeneic blood transfusion are major complications of cardiac surgery, which increase perioperative complications, perioperative mortality and medical costs. This study addresses the unmet need for optimizing coagulation management in cardiac surgery by comparing the efficacy and safety of 4-factor prothrombin complex concentrates (PCC) and fresh frozen plasma (FFP). he trial is designed as a non-inferiority, randomized controlled study to assess whether PCC is non-inferior to FFP in reducing perioperative blood loss and transfusion needs in patients undergoing cardiac surgery with cardiopulmonary bypass (CPB). Patients who signed informed consent, aged 18 to 80 years, receiving elective CABG or valve replacement or valvuloplasty under CPB will be included. 816 subjects will be randomly divided into 2 groups (PCC group and FFP group), with 408 cases in each group. Preoperative management, anesthetic and surgical techniques will be standardized for both groups. When activated partial thromboplastin time (APTT) is prolonged (> 45 s), patients will be given 8~15 IU/kg PCC or 6~10 ml/kg FFP according to the allocation. All the patients will be followed up respectively at 24 hours, 48 hours, 72 hours and 7 days after the surgery to record observations relevant to the study and the results of laboratory testing. The laboratory tests include hemoglobin concentration, hematocrit, platelet count, INR, PT, APTT, fibrinogen levels and blood biochemistry parameters. The primary outcome is the volume of blood loss within 24 hours after surgery. The secondary outcomes include (1) the total units of allogeneic red blood cells (RBCs) transfused within 7 days after surgery and (2) hemostatic response (effective if no hemostatic interventions occurred from 60 minutes to 24 hours after treatment initiation). Adverse events and serious adverse events will be monitored as safety outcomes.

Modified intent-to-treat analysis will be used for all valid variables. All randomised subjects in the study, regardless of adherence to the study process or whether an adverse event occurs before or after the intervention, should be included in the analysis. Sensitivity analysis will be performed to assess potential bias from protocol deviations or missing data. Baseline characteristics will be tabulated and compared between the PCC and FFP groups using absolute standardised differences, and the threshold will be calculated using the formula (1.96×√[n1+n2]/[n1×n2]). A value exceeding this threshold will be considered imbalanced between groups. Unbalanced baseline factors and different study centers will be further adjusted by multivariable regression models.

The primary outcome, the volume of blood loss within 24 hours after surgery, will be compared using one-tailed ttest. If there exists unbalanced baseline characteristics, the treatment effect (difference in means between the PCC and FFP groups) will be estimated using a linear regression model adjusted for centers and any imbalanced baseline covariates. The non-inferiority test will be conducted using the estimated difference minus the non-inferiority margin (200 mL) in the numerator, and the estimated standard error of the difference in the denominator. Non-inferiority will be concluded if the upper bound of the 99.7% confidence interval was below the predefined non-inferiority margin of 200 mL, corresponding to a one-sided P value < 0.025. For the continuous secondary outcome, the total units of allogeneic RBCs transfused during and within 7 days after surgery will be compared using a t-test with log transformation of the variable. The rate of hemostatic response will be compared using the chi-square test. Treatment effects will be reported as risk ratios and mean differences for binary and continuous outcomes respectively with 95% confidence intervals. If there exists unbalanced baseline characteristics, the secondary outcomes will be regressed against the group allocation, centers and the unbalanced factors using linear regression or Poisson regression models. The following subgroups will be analysed: age (<65 years/ ≥65 years), gender (male/female), study center, NYHA class (I and II/III and IV), surgery type (simple/complex surgery) and CPB duration (≤120 minutes, 121-180 minutes, >180 minutes). For safety outcomes, we will only describe the incidence of overall adverse events, SAEs, and component adverse events without statistical tests between two groups. A two-sided P-value < 0.05 was considered indicative of statistical significance.

Our independent Data Safety Monitoring Board (DSMB), which includes an epidemiologist, a pharmacologist, an anesthesiologist, and a blood transfusion specialist, conducted an interim review of our study. Considering the shortage of blood resources and the difficulties in large-sample recruitment, the DSMB recommended adding an interim analysis. Therefore, an interim analysis was planned after 50% of the target enrollment had been achieved. o ensure statistical rigor, the Lan-DeMets alpha-spending approach with O'Brien-Fleming boundaries was implemented for interim efficacy and futility evaluation, offering conservative thresholds early in the trial. With the same standard deviation (824.38 mL) and the superior margin (200 mL) is, as well as the 90% power and 10% dropout rate, we recalculated the sample size and found out that 816 patients in total should be recruited. Thus our interim analysis will be conducted when 408 patients recruited.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years.
2. Undergoing elective coronary artery bypass grafting (CABG) or valve replacement or valvuloplasty through CPB.
3. Signing of the informed consent form.
4. Developing coagulation factor deficiency or coagulopathic bleeding during the surgery, meeting the indications of PCC or FFP treatment: a) prolonged APTT (> 45 s) measured 20 minutes after CPB, and b) excessive bleeding observed.

Exclusion Criteria:

1. History of cardiac surgery.
2. Severe hepatic dysfunction before surgery.
3. Coagulopathy before surgery, including inherited or acquired coagulation factor deficiencies, thrombocytopenia, platelet dysfunction and other bleeding disorders.
4. Use of warfarin and INR > 1.2 before surgery.
5. Withdrawal of clopidogrel less than 5 days and low molecular weight heparin less than 12 hours before surgery.
6. Allergy to allogeneic blood products.
7. Pregnancy.
8. Other serious diseases that may affect patient survival time, such as cancers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 820 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
volume of blood loss within 24 hours after surgery | postoperative period up to 24 hours after surgery
  the volume of drainage within 24 hours after surgery

SECONDARY OUTCOMES:
total units of allogeneic RBCs transfused within 7 days after surgery | during the intraoperative and postoperative period up to 7 days after surgery
  the total units of allogeneic RBC transfused during the intraoperative and postoperative the total units of allogeneic RBCs transfused during and within 7 days after surgery
hemostatic response | from 60 minutes to 24 hours after treatment initiation
  effective if no hemostatic interventions occurred from 60 minutes to 24 hours after treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Lijian Pei, M.D., Study Chair — Peking Union Medical College Hospital; Jia Shi, M.D., Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (2):
- China (2):
  - Cardiovascular Institute and Fuwai Hospital, CAMS&PUMC, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Yes
Specific IPD could be obtained from Lijian Pei (hazelbeijing@vip.163.com).
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Parr KG, Patel MA, Dekker R, Levin R, Glynn R, Avorn J, Morse DS. Multivariate predictors of blood product use in cardiac surgery. J Cardiothorac Vasc Anesth. 2003 Apr;17(2):176-81. doi: 10.1053/jcan.2003.44. PMID 12698398
- [Background] Moulton MJ, Creswell LL, Mackey ME, Cox JL, Rosenbloom M. Reexploration for bleeding is a risk factor for adverse outcomes after cardiac operations. J Thorac Cardiovasc Surg. 1996 May;111(5):1037-46. doi: 10.1016/s0022-5223(96)70380-x. PMID 8622301
- [Background] Mariscalco G, Biancari F, Juvonen T, Zanobini M, Cottini M, Banach M, Murphy GJ, Beghi C, Angelini GD. Red blood cell transfusion is a determinant of neurological complications after cardiac surgery. Interact Cardiovasc Thorac Surg. 2015 Feb;20(2):166-71. doi: 10.1093/icvts/ivu360. Epub 2014 Nov 2. PMID 25368133
- [Background] Alfirevic A, Xu M, Johnston D, Figueroa P, Koch CG. Transfusion increases the risk for vasoplegia after cardiac operations. Ann Thorac Surg. 2011 Sep;92(3):812-9. doi: 10.1016/j.athoracsur.2011.04.020. Epub 2011 Jul 23. PMID 21788009
- [Background] Sellman M, Intonti MA, Ivert T. Reoperations for bleeding after coronary artery bypass procedures during 25 years. Eur J Cardiothorac Surg. 1997 Mar;11(3):521-7. doi: 10.1016/s1010-7940(96)01111-6. PMID 9105818
- [Background] Ottino G, De Paulis R, Pansini S, Rocca G, Tallone MV, Comoglio C, Costa P, Orzan F, Morea M. Major sternal wound infection after open-heart surgery: a multivariate analysis of risk factors in 2,579 consecutive operative procedures. Ann Thorac Surg. 1987 Aug;44(2):173-9. doi: 10.1016/s0003-4975(10)62035-8. PMID 3619541
- [Background] Zacharias A, Habib RH. Factors predisposing to median sternotomy complications. Deep vs superficial infection. Chest. 1996 Nov;110(5):1173-8. doi: 10.1378/chest.110.5.1173. PMID 8915216
- [Background] Linden MD. The hemostatic defect of cardiopulmonary bypass. J Thromb Thrombolysis. 2003 Dec;16(3):129-47. doi: 10.1023/B:THRO.0000024051.12177.e9. PMID 15087599
- [Background] Society of Thoracic Surgeons Blood Conservation Guideline Task Force; Ferraris VA, Ferraris SP, Saha SP, Hessel EA 2nd, Haan CK, Royston BD, Bridges CR, Higgins RS, Despotis G, Brown JR; Society of Cardiovascular Anesthesiologists Special Task Force on Blood Transfusion; Spiess BD, Shore-Lesserson L, Stafford-Smith M, Mazer CD, Bennett-Guerrero E, Hill SE, Body S. Perioperative blood transfusion and blood conservation in cardiac surgery: the Society of Thoracic Surgeons and The Society of Cardiovascular Anesthesiologists clinical practice guideline. Ann Thorac Surg. 2007 May;83(5 Suppl):S27-86. doi: 10.1016/j.athoracsur.2007.02.099. PMID 17462454
- [Background] Dacey LJ, Munoz JJ, Baribeau YR, Johnson ER, Lahey SJ, Leavitt BJ, Quinn RD, Nugent WC, Birkmeyer JD, O'Connor GT. Reexploration for hemorrhage following coronary artery bypass grafting: incidence and risk factors. Northern New England Cardiovascular Disease Study Group. Arch Surg. 1998 Apr;133(4):442-7. doi: 10.1001/archsurg.133.4.442. PMID 9565127
- [Background] Despotis G, Eby C, Lublin DM. A review of transfusion risks and optimal management of perioperative bleeding with cardiac surgery. Transfusion. 2008 Mar;48(1 Suppl):2S-30S. doi: 10.1111/j.1537-2995.2007.01573.x. No abstract available. PMID 18302579
- [Background] Karkouti K, Callum J, Crowther MA, McCluskey SA, Pendergrast J, Tait G, Yau TM, Beattie WS. The relationship between fibrinogen levels after cardiopulmonary bypass and large volume red cell transfusion in cardiac surgery: an observational study. Anesth Analg. 2013 Jul;117(1):14-22. doi: 10.1213/ANE.0b013e318292efa4. Epub 2013 May 17. PMID 23687229
- [Background] Weber CF, Klages M, Zacharowski K. Perioperative coagulation management during cardiac surgery. Curr Opin Anaesthesiol. 2013 Feb;26(1):60-4. doi: 10.1097/ACO.0b013e32835afd28. PMID 23222215
- [Background] Khuri SF MA, Valeri CR. The effects of cardiopulmonary bypass on hemostasis. Loscabo J, Schafer AI, eds. Thrombosis & Hemorrhage. Cambridge: Blackwell Science. 1993;1993:1051-1073.
- [Background] Kaspereit F, Hoffmann S, Pragst I, Dickneite G. Prothrombin complex concentrate mitigates diffuse bleeding after cardiopulmonary bypass in a porcine model. Br J Anaesth. 2010 Nov;105(5):576-82. doi: 10.1093/bja/aeq216. Epub 2010 Aug 17. PMID 20716565
- [Background] Stanworth SJ, Brunskill SJ, Hyde CJ, McClelland DB, Murphy MF. Is fresh frozen plasma clinically effective? A systematic review of randomized controlled trials. Br J Haematol. 2004 Jul;126(1):139-52. doi: 10.1111/j.1365-2141.2004.04973.x. PMID 15198745
- [Background] Sun JC, Davidson MJ, Lamy A, Eikelboom JW. Antithrombotic management of patients with prosthetic heart valves: current evidence and future trends. Lancet. 2009 Aug 15;374(9689):565-76. doi: 10.1016/S0140-6736(09)60780-7. PMID 19683642
- [Background] Eitz T, Schenk S, Fritzsche D, Bairaktaris A, Wagner O, Koertke H, Koerfer R. International normalized ratio self-management lowers the risk of thromboembolic events after prosthetic heart valve replacement. Ann Thorac Surg. 2008 Mar;85(3):949-54; discussion 955. doi: 10.1016/j.athoracsur.2007.08.071. PMID 18291177
- [Background] Safaoui MN, Aazami R, Hotz H, Wilson MT, Margulies DR. A promising new alternative for the rapid reversal of warfarin coagulopathy in traumatic intracranial hemorrhage. Am J Surg. 2009 Jun;197(6):785-90. doi: 10.1016/j.amjsurg.2008.04.003. Epub 2008 Aug 22. PMID 18722586
- [Background] Fariborz Farsad B, Golpira R, Najafi H, Totonchi Z, Salajegheh S, Bakhshandeh H, Hashemian F. Comparison between Prothrombin Complex Concentrate (PCC) and Fresh Frozen Plasma (FFP) for the Urgent Reversal of Warfarin in Patients with Mechanical Heart Valves in a Tertiary Care Cardiac Center. Iran J Pharm Res. 2015 Summer;14(3):877-85. PMID 26330876
- [Background] Cromwell C, Aledort LM. FEIBA: a prohemostatic agent. Semin Thromb Hemost. 2012 Apr;38(3):265-7. doi: 10.1055/s-0032-1309286. Epub 2012 Mar 29. PMID 22460908
- [Background] Franchini M, Lippi G. Prothrombin complex concentrates: an update. Blood Transfus. 2010 Jul;8(3):149-54. doi: 10.2450/2010.0149-09. No abstract available. PMID 20671873
- [Background] Hellstern P. Production and composition of prothrombin complex concentrates: correlation between composition and therapeutic efficiency. Thromb Res. 1999 Aug 15;95(4 Suppl 1):S7-12. doi: 10.1016/s0049-3848(99)00078-x. PMID 10499903
- [Background] Cappabianca G, Mariscalco G, Biancari F, Maselli D, Papesso F, Cottini M, Crosta S, Banescu S, Ahmed AB, Beghi C. Safety and efficacy of prothrombin complex concentrate as first-line treatment in bleeding after cardiac surgery. Crit Care. 2016 Jan 6;20:5. doi: 10.1186/s13054-015-1172-6. PMID 26738468
- [Background] Song HK, Tibayan FA, Kahl EA, Sera VA, Slater MS, Deloughery TG, Scanlan MM. Safety and efficacy of prothrombin complex concentrates for the treatment of coagulopathy after cardiac surgery. J Thorac Cardiovasc Surg. 2014 Mar;147(3):1036-40. doi: 10.1016/j.jtcvs.2013.11.020. Epub 2013 Dec 22. PMID 24365268
- [Background] Weinberger J, Cipolle M. Optimal Reversal of Novel Anticoagulants in Trauma. Crit Care Clin. 2017 Jan;33(1):135-152. doi: 10.1016/j.ccc.2016.08.005. PMID 27894493
- [Background] Ortmann E, Besser MW, Sharples LD, Gerrard C, Berman M, Jenkins DP, Klein AA. An exploratory cohort study comparing prothrombin complex concentrate and fresh frozen plasma for the treatment of coagulopathy after complex cardiac surgery. Anesth Analg. 2015 Jul;121(1):26-33. doi: 10.1213/ANE.0000000000000689. PMID 25822921
- [Background] Patanwala AE, Acquisto NM, Erstad BL. Prothrombin complex concentrate for critical bleeding. Ann Pharmacother. 2011 Jul;45(7-8):990-9. doi: 10.1345/aph.1Q096. Epub 2011 Jul 5. PMID 21730276
- [Background] Hellstern P, Halbmayer WM, Kohler M, Seitz R, Muller-Berghaus G. Prothrombin complex concentrates: indications, contraindications, and risks: a task force summary. Thromb Res. 1999 Aug 15;95(4 Suppl 1):S3-6. doi: 10.1016/s0049-3848(99)00077-8. No abstract available. PMID 10499902
- [Background] Huttner HB, Schellinger PD, Hartmann M, Kohrmann M, Juettler E, Wikner J, Mueller S, Meyding-Lamade U, Strobl R, Mansmann U, Schwab S, Steiner T. Hematoma growth and outcome in treated neurocritical care patients with intracerebral hemorrhage related to oral anticoagulant therapy: comparison of acute treatment strategies using vitamin K, fresh frozen plasma, and prothrombin complex concentrates. Stroke. 2006 Jun;37(6):1465-70. doi: 10.1161/01.STR.0000221786.81354.d6. Epub 2006 May 4. PMID 16675739
- [Background] Erber WN, Perry DJ. Plasma and plasma products in the treatment of massive haemorrhage. Best Pract Res Clin Haematol. 2006;19(1):97-112. doi: 10.1016/j.beha.2005.01.026. PMID 16377544
- [Background] Vigue B, Ract C, Tremey B, Engrand N, Leblanc PE, Decaux A, Martin L, Benhamou D. Ultra-rapid management of oral anticoagulant therapy-related surgical intracranial hemorrhage. Intensive Care Med. 2007 Apr;33(4):721-5. doi: 10.1007/s00134-007-0528-z. Epub 2007 Jan 27. PMID 17260127
- [Background] Levy JH, Tanaka KA, Dietrich W. Perioperative hemostatic management of patients treated with vitamin K antagonists. Anesthesiology. 2008 Nov;109(5):918-26. doi: 10.1097/ALN.0b013e3181895bd8. PMID 18946305
- [Background] Leissinger CA, Blatt PM, Hoots WK, Ewenstein B. Role of prothrombin complex concentrates in reversing warfarin anticoagulation: a review of the literature. Am J Hematol. 2008 Feb;83(2):137-43. doi: 10.1002/ajh.21046. PMID 17729241
- [Background] Bux J. Transfusion-related acute lung injury (TRALI): a serious adverse event of blood transfusion. Vox Sang. 2005 Jul;89(1):1-10. doi: 10.1111/j.1423-0410.2005.00648.x. PMID 15938734
- [Background] Ansell J, Hirsh J, Hylek E, Jacobson A, Crowther M, Palareti G. Pharmacology and management of the vitamin K antagonists: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines (8th Edition). Chest. 2008 Jun;133(6 Suppl):160S-198S. doi: 10.1378/chest.08-0670. PMID 18574265
- [Background] Pabinger I, Brenner B, Kalina U, Knaub S, Nagy A, Ostermann H; Beriplex P/N Anticoagulation Reversal Study Group. Prothrombin complex concentrate (Beriplex P/N) for emergency anticoagulation reversal: a prospective multinational clinical trial. J Thromb Haemost. 2008 Apr;6(4):622-31. doi: 10.1111/j.1538-7836.2008.02904.x. Epub 2008 Jan 15. PMID 18208533
- [Background] Pabinger-Fasching I. Warfarin-reversal: results of a phase III study with pasteurised, nanofiltrated prothrombin complex concentrate. Thromb Res. 2008;122 Suppl 2:S19-22. doi: 10.1016/S0049-3848(08)70005-7. PMID 18549908
- [Background] Nienaber U, Innerhofer P, Westermann I, Schochl H, Attal R, Breitkopf R, Maegele M. The impact of fresh frozen plasma vs coagulation factor concentrates on morbidity and mortality in trauma-associated haemorrhage and massive transfusion. Injury. 2011 Jul;42(7):697-701. doi: 10.1016/j.injury.2010.12.015. Epub 2011 Mar 9. PMID 21392760
- [Background] Goldstein JN, Refaai MA, Milling TJ Jr, Lewis B, Goldberg-Alberts R, Hug BA, Sarode R. Four-factor prothrombin complex concentrate versus plasma for rapid vitamin K antagonist reversal in patients needing urgent surgical or invasive interventions: a phase 3b, open-label, non-inferiority, randomised trial. Lancet. 2015 May 23;385(9982):2077-87. doi: 10.1016/S0140-6736(14)61685-8. Epub 2015 Feb 27. PMID 25728933
- [Background] Green L, Roberts N, Cooper J, Field J, Gill R, Klein A, Agarwal S, Stanworth S, Johnston A, Monk V, O'Brien B. A pragmatic pilot phase II randomised controlled trial of prothrombin complex concentrates (PCC) versus fresh frozen plasma (FFP) in adult patients who are undergoing heart surgery (PROPHESY). Trials. 2019 Dec 9;20(1):684. doi: 10.1186/s13063-019-3759-8. PMID 31815658
- [Background] Kozek-Langenecker SA, Afshari A, Albaladejo P, Santullano CA, De Robertis E, Filipescu DC, Fries D, Gorlinger K, Haas T, Imberger G, Jacob M, Lance M, Llau J, Mallett S, Meier J, Rahe-Meyer N, Samama CM, Smith A, Solomon C, Van der Linden P, Wikkelso AJ, Wouters P, Wyffels P. Management of severe perioperative bleeding: guidelines from the European Society of Anaesthesiology. Eur J Anaesthesiol. 2013 Jun;30(6):270-382. doi: 10.1097/EJA.0b013e32835f4d5b. PMID 23656742
- [Derived] Hayes K, Fernando MC, Jordan V. Prothrombin complex concentrate in cardiac surgery for the treatment of coagulopathic bleeding. Cochrane Database Syst Rev. 2022 Nov 21;11(11):CD013551. doi: 10.1002/14651858.CD013551.pub2. PMID 36408876
- [Derived] Pei L, Sun C, Lv H, Zhang Y, Shi J. Efficacy of prothrombin complex concentrate (PCC) versus fresh frozen plasma (FFP) in reducing perioperative blood loss in cardiac surgery: study protocol for a non-inferiority, randomised controlled trial. BMJ Open. 2022 Feb 10;12(2):e051072. doi: 10.1136/bmjopen-2021-051072. PMID 35144945